CLINICAL TRIAL: NCT05335057
Title: Effects of Social Presence and Perception on Pain: Comparing Close Others to Strangers and VR to Video Conferencing
Brief Title: Effects of Social Presence and Perception in Virtual Reality on Pain (SPP)
Acronym: SPP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1701006910-2
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Pain Threshold
Keywords: virtual reality

STUDY DESIGN:
Intervention Model Description: Each participant will experience all four conditions, in a random order
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Time 1 (Active Comparator): Participant will be randomly assigned to one of the four interventions; either Near Non-Social, Near Social, Far Non-Social, or Far Social
  Interventions: Behavioral: VR Close Other; Behavioral: VR Alone; Behavioral: VR Stranger; Behavioral: Video Close Other
- Time 2 (Active Comparator): Participant will be randomly assigned to one of the remaining three interventions; either Near Non-Social, Near Social, Far Non-Social, or Far Social
  Interventions: Behavioral: VR Close Other; Behavioral: VR Alone; Behavioral: VR Stranger; Behavioral: Video Close Other
- Time 3 (Active Comparator): Participant will be randomly assigned to one of the remaining two interventions; either Near Non-Social, Near Social, Far Non-Social, or Far Social
  Interventions: Behavioral: VR Close Other; Behavioral: VR Alone; Behavioral: VR Stranger; Behavioral: Video Close Other
- Time 4 (Experimental): Participant will be randomly assigned to the remainingintervention; either Near Non-Social, Near Social, Far Non-Social, or Far Social
  Interventions: Behavioral: VR Close Other; Behavioral: VR Alone; Behavioral: VR Stranger; Behavioral: Video Close Other

INTERVENTIONS:
Behavioral: VR Close Other — Participants will be stably seated, and observed by a research assistant, as they complete an induced pain threshold task while they experience one of four randomly assigned virtual environments while chatting with the friend or family member who accompanied them to the lab
Behavioral: VR Alone — Participants will be stably seated, and observed by a research assistant, as they complete an induced pain threshold task while they experience one of four randomly assigned virtual environments alone
Behavioral: VR Stranger — Participants will be stably seated, and observed by a research assistant, as they complete an induced pain threshold task while they experience one of four randomly assigned virtual environments while chatting with a stranger
Behavioral: Video Close Other — Participants will be stably seated, and observed by a research assistant, as they complete an induced pain threshold task while they chat with the friend or family member who accompanied them to the lab using a video-conferencing tool

SUMMARY:
This experiment aims to examine the effects of social interaction with close others or strangers in virtual reality or through a video-conferencing call, on pain threshold in healthy volunteers in an induced pain task.

In a within-subjects study, participants will complete a series of induced-pain heat ramps in four conditions. These conditions are 1. alone in virtual reality 2. with a close friend or family member in virtual reality 3. with a stranger in virtual reality 4. with the same close friend or family member in a video call.

DETAILED DESCRIPTION:
Some of the earliest clinical uses of virtual reality were as a distractor for patients experiencing pain. However, virtual worlds also allow for social interaction, which has the potential to strongly affect both pain and the sensation of presence in an environment. While social support has been linked to pain reduction, in a recent study, participants who texted with a stranger while undergoing surgery were less likely to require analgesia than those who texted with companions or played a distracting game on their phone. While the authors propose that the context of the chat may have affected participants' pain levels, another additive possibility is that these patients were experiencing social presence with the strangers, who were conversing from a location outside the hospital, and were thus feeling less present in the hospital environment. This might explain why participants received greater benefit from these text conversations than from conversations with loved ones, who were conversing from the hospital environment where their pain occurred. In a previous study, we found that participants in an induced pain task demonstrated higher pain thresholds when they were interacting socially with a stranger compared to when they were alone (Won, Pandita and Kruzan, 2020).

In this study, we follow up on these results. First, we aim to replicate the previous finding of social interactions, overall, increasing pain tolerance. Second, we aim to compare the potential effects of interacting with a stranger compared to a "close other," defined as a friend or family member. Third, we compare social interactions in virtual reality compared to video. Fourth, we examine whether cortisol is linked with pain threshold.

METHODS AND RESEARCH STRATEGY: Our previous study used 75 participants, and since this is the closest study to our current research design, we will retain this number as our target. We will work with a student sample of convenience.

Each participant will experience four conditions in a random order: 1. alone in virtual reality 2. with a close friend or family member in virtual reality 3. with a stranger in virtual reality 4. with the same close friend or family member in a video call. Each condition will take place in a different virtual environment.

Participants will be stably seated, and observed by a research assistant, as they experience each condition. During each condition, participants will complete an induced pain task using a Medoc TSA-2001/Model Q-Sense thermode. Prior to experiencing the four experimental conditions, participants will complete a "practice" induced pain task while viewing a different virtual environment. This will allow them to orient themselves to both the virtual environment and the pain task, since based on the pilot experiment, order effects are predicted to be most notable for the first pain task administered. In this and all subsequent induced pain tasks, participants will place their non-dominant hand on the thermode and will be instructed to remove their hand as soon as they feel the temperature has become "painful". The beginning and end of each trial (when the heat ramp begins, and when participants remove their hands) will be noted, and that time duration, and thus the degree of temperature to which it corresponds, will serve as the measure of pain threshold for that trial. In addition to this outcome measure, after each pain trial participants will also fill out a brief self-report survey. These measures will include their self-reported feelings of presence in the virtual environment, and social presence with the other conversational partners. All conditions will be presented in a randomized order to control for order effects. The time to complete these surveys will be approximately 7-10 minutes, which will also allow participants time between each trial to reorient themselves to the real environment, and for any lingering effects of heat on their hands to dissipate. After each survey, 15 minutes after each pain task, a saliva sample for cortisol will be taken.

ELIGIBILITY:
Inclusion Criteria:

Consenting Adult

Exclusion Criteria:

1. History of cardiovascular disorder
2. History of fainting or seizures
3. Open cut or sore on hand to be thermally tested
4. Burn or sunburn on hand to be thermally tested.
5. Pregnancy
6. Prone to motion sickness, or have balance or dizziness conditions
7. Recent concussion
8. Seizure disorders
9. History of fainting or seizures
10. Visual impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Pain threshold in degrees tolerated at end of trial | The beginning and end of each trial < 90 seconds
  Change in temperature from the beginning to the end of each trial (when the heat ramp begins, and when participants remove their hands) will be noted in milliseconds.

SECONDARY OUTCOMES:
Cortisol levels | 15 minutes between samples
  Cortisol levels derived from saliva samples
Self-reported Social Presence | Experience and subsequent survey time 5-15 minutes
  Questionnaire of self-reported feelings of social presence with the conversational partner (1-5 Likert scale, higher means greater)
Self-reported Environmental Presence | Experience and subsequent survey time 5-15 minutes
  Questionnaire of self-reported feelings of environmental presence with the conversational partner (1-5 Likert scale, higher means greater)

CONTACTS AND LOCATIONS:
Locations (1):
- Cornell Virtual Embodiment Lab, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and code will be posted through the Cornell Center for Social Sciences and Cornell Restricted Access Data Center repositories after publication and made available to researchers who present a valid IRB protocol and promise to destroy data after use.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The SAP is already posted to Open Science Framework. Once published the data will be available on the CCSS/CRADC archives indefinitely.
Access Criteria: Anonymized data will be available to any who request it. The full data set will be available upon submission of a valid IRB protocol and promise to destroy data after use.